CLINICAL TRIAL: NCT06946862
Title: Investigation of Factors Influencing Treatment Expectations in Individuals With Chronic Neck Pain
Brief Title: Factors Affecting Treatment Expectations in Chronic Neck Pain
Status: Completed | Type: Observational
Sponsor: KTO Karatay University (Other)
Responsible Party: Sponsor
Other Study IDs: KaratayUBD2
Record Dates: First submitted 2025-04-21; First posted 2025-04-27 (Actual); Last update posted 2025-08-06 (Actual); Status verified 2025-04

CONDITIONS: Neck Pain Chronic
MeSH Terms: interventions — Dosage Forms; Methods

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Cohort1-Chronic Neck Pain Group: Participants in this cohort are adults diagnosed with chronic neck pain lasting longer than three months. They may experience nonspecific mechanical or postural neck pain without any specific underlying pathology. Individuals with chronic neck pain of varying severity levels who meet the inclusion criteria are included in this group.
  Interventions: Other: no treatment, medication or intervention

INTERVENTIONS:
Other: no treatment, medication or intervention — will make an observational assessment of the participants' treatment expectations. Participants will not be subjected to any treatment or intervention, only their current situation will be observed.

SUMMARY:
The aim of this study was to determine which factors affect treatment expectations in individuals with chronic neck pain.

DETAILED DESCRIPTION:
This study aims to investigate the factors that influence treatment expectations in individuals with chronic neck pain.

Neck pain is one of the most common musculoskeletal conditions and a major public health issue that significantly affects quality of life and imposes economic burdens due to healthcare costs and productivity loss. It is considered the fourth leading cause of disability worldwide. Chronic neck pain is increasingly prevalent due to modern lifestyle factors, such as prolonged use of smartphones and computers, and is most often classified as nonspecific, mechanical, or postural in origin.

Numerous biopsychosocial factors have been associated with the onset and persistence of neck pain, including age, gender, occupation, duration of sitting or sedentary work, smoking, stress, anxiety, depression, personality traits, emotional state, and levels of physical activity.

Treatment expectations are a key determinant of treatment response and clinical outcomes in musculoskeletal disorders. Positive expectations have been shown to enhance treatment effects, while negative expectations (nocebo effects) may worsen outcomes. Understanding these expectations may aid in tailoring treatment approaches and improving communication between patients and healthcare providers.

This study will evaluate demographic, psychological, and behavioral factors that may influence the treatment expectations of patients with chronic neck pain. The findings may contribute to improving treatment planning, patient education, and shared decision-making in clinical practice.

ELIGIBILITY:
Inclusion Criteria:

* Having been diagnosed with chronic neck pain by a Physical Medicine and Rehabilitation Specialist
* Being between 18 and 80 years of age
* Signing a consent form after receiving verbal information

Exclusion Criteria:

* Presence of instability in the neck joints
* Trauma within the last year
* Advanced osteoporosis
* Previous neck surgery
* Physical therapy within the last 6 months
* Neurological findings or radiculopathy

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: neck pain chronic
Sampling Method: Probability Sample
Enrollment: 100 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-07-01 (Actual); Study Completion 2025-08-01 (Actual)

PRIMARY OUTCOMES:
Treatment Expectation Questionnaire | Baseline
  Developed by Shedden-Mora et al. (2023) (15), it is a psychological assessment tool used to measure patients' expectations about treatment before starting a treatment process. The Turkish validity and reliability study of the questionnaire was conducted by Çakır et al. (2024) (24). Validity Measurements The main items of the questionnaire, which consists of 15 main items and 6 additional questions, are structured as a scale in which the patient marks his/her expectation between 0 and 10. The questionnaire consists of treatment benefit (items 1-3), positive effect (items 4-6), negative events (items 7-9), negative effect (items 10-11), process (items 12-13) and behaviour control (items 14-15) subscales.

SECONDARY OUTCOMES:
Pain Beliefs Scale | Baseline
  It was developed by Edwards et al. (1992) to evaluate beliefs about the cause and treatment of pain (25). The Turkish validity and reliability study of the questionnaire was conducted by Berk (2006). The scale has a total of 12 items and consists of two test domains: 8-item Organic Beliefs and 4-item Psychological Beliefs. Participants are asked to tick the most appropriate one for themselves from 6 options ranging from 1. 'never' to 6. 'always'. Each item is given a score between 1 and 6, and the score of each subtest is calculated by averaging the scores of the items belonging to that subtest. There is no cut-off point for the scale and high scores indicate high pain beliefs and low scores indicate low pain beliefs. The highest score for organic and psychological beliefs is 6 and the lowest score is 1.
Pain Self-Efficacy Questionnaire | Baseline
  It is a questionnaire developed by Michael K. Nicholas (1989), consisting of 10 items, easy to understand, can be applied without taking time, evaluates the role of pain in establishing social relationships, doing hobbies or housework, and questions the use of analgesics in coping with pain. The Turkish validity and reliability study of the questionnaire was conducted by Doğan (2019). Individuals with chronic pain are asked to score how safely they can perform the defined activities despite their pain. Scoring is done on a 7-point Likert scale, where 0 = 'completely unsafe' and 6 = 'completely safe'. By summing the scores of 10 items, a high score indicates a strong self-efficacy belief according to the total score between 0 and 60.
Hospital Anxiety and Depression Scale | Baseline
  It was developed by Zigmond and Snaith (1983) to determine the risk of anxiety and depression and to measure the level and change in severity. The Turkish validity and reliability study of the scale was conducted by Aydemir et al. (1997) (30). It consists of 14 items, 7 of which investigate symptoms of depression and 7 of which investigate symptoms of anxiety. Odd numbers measure anxiety and even numbers measure depression. Responses are evaluated in a 4-point Likert scale and scored between 0-3. Patients score between 0 and 21 on both subscales. The cut-off points of the Turkish form of the HADÖ were determined as 10 for the anxiety subscale and 7 for the depression subscale. Scores above these values are considered as risk for depression and anxiety.
Visual Analogue Scale | Baseline
  It is a scale developed by Price et al. (1983) to measure the severity of pain in individuals. The scale consists of a 10 cm horizontally positioned line on the page. The number '0', which is the starting point on this line, represents that the patient does not feel any pain, and the number '10' represents the worst pain experienced by the patient within his/her own experience. The patient is asked to mark anywhere on this straight line between 0 and 10 to indicate the pain he/she had at the time the test was administered. Then, with the help of a ruler, the distance of the point marked by the patient to the starting point, the number 0, is measured in cm and the intensity of the pain is determined.

CONTACTS AND LOCATIONS:
Overall Officials: Burcu DURSUN, Lecturer, Principal Investigator — KTO Karatay University
Locations (1):
- Kto Karatay Üniversitesi, Karatay, Konya, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participant data from this study will be shared upon reasonable request after the completion and publication of the study results. All data will be anonymized to ensure participant confidentiality and privacy. Data sharing will be subject to approval by the study investigators and may require a data use agreement to protect sensitive information.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Data will be retained and available for sharing for 5 years following the completion of the study.
Access Criteria: Access to de-identified individual participant data will be granted to qualified researchers who submit a reasonable request detailing the purpose and methods of their proposed analysis. Approval from the study investigators is required prior to data release. Researchers must agree to maintain confidentiality and use the data solely for scientific research purposes. A data use agreement will be signed to ensure responsible handling of the information.